CLINICAL TRIAL: NCT00142779
Title: Serotonin Treatment of Cocaine Dependence
Brief Title: Fluoxetine to Reduce Cocaine Use in Cocaine and Opioid Addicts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Eric C. Strain, Johns Hopkins University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-10754-2; R01-10754-2; DPMC
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2009-05

CONDITIONS: Cocaine-Related Disorders; Opioid-Related Disorders
Keywords: Cocaine Addiction; Cocaine Dependence; Opiate Addiction; Opiate Dependence
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders | interventions — Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine

SUMMARY:
Cocaine addiction is a serious health problem with no available medical treatment for preventing relapse. Fluoxetine, a medication that is currently used to treat depression and anxiety disorders, may also be effective at diminishing cocaine use in individuals with severe cocaine addiction. This study will evaluate the effectiveness of fluoxetine at reducing cocaine use in individuals addicted to cocaine and opioids who are concurrently receiving methadone treatment.

DETAILED DESCRIPTION:
Individuals addicted to cocaine often experience feelings of restlessness, irritability, anxiety, and paranoia. Reducing cocaine use can lead to depression. In an attempt to alleviate the depressive symptoms, individuals may resume drug use. Fluoxetine, a medication that is currently used to treat depression and panic attacks, may assist at reducing cocaine use in individuals addicted to cocaine. By increasing serotonin, a chemical in the brain that helps maintain mental balance, fluoxetine may lessen depressive symptoms and decrease the reinforcing effects of cocaine. Voucher incentive programs, in which items or services are offered as a reward for remaining drug-free, are also a useful component of substance abuse treatment. Preliminary research has shown that fluoxetine, when combined with an incentive program, is an effective treatment for reducing cocaine use. Further research is needed to confirm the benefits of fluoxetine for cocaine and opioid addicts. The purpose of this study is to evaluate the effectiveness of fluoxetine, in combination with a voucher incentive program, at reducing cocaine use in methadone-maintained cocaine and opioid addicts.

This 33-week study will enroll individuals addicted to both cocaine and opioids who are concurrently enrolled in a methadone treatment program. Participants will be randomly assigned to receive either 60 mg of fluoxetine or placebo on a daily basis for 12 weeks from Weeks 8 through 19. Study visits will occur once a week. Questionnaires and self-reports will be completed to assess medication side effects and cocaine use. Cocaine levels will be monitored three times a week with urine tests. During the 12 weeks of treatment, participants will also be randomly assigned to either take part in a voucher incentives program or not take part in the program. Participants in the voucher program will receive a voucher that may be exchanged for various items and services for each urine test with a negative cocaine result.

ELIGIBILITY:
Inclusion Criteria:

* Currently dependent on opioids
* Currently dependent on cocaine
* Eligible to receive methadone maintenance treatment

Exclusion Criteria:

* Current significant medical or psychiatric illness
* Current use of a specific serotonin reuptake inhibitor (SSRI)
* History of allergy to SSRI medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220
Dates: Start 2001-04; Primary Completion 2006-01 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Cocaine use (measured by urine screen and self-report at Week 19 and 33)
Medication side effects (measured by self-reports throughout Weeks 8 through 19)

CONTACTS AND LOCATIONS:
Overall Officials: Eric C. Strain, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States